CLINICAL TRIAL: NCT06661395
Title: Adaption of the Wingate Test to Virtual Reality Based Wearable Technology
Brief Title: Integration of the Wingate Test Into Virtual Reality Based System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gizem yilmaz, Research Assisstant, Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: E-10840098-772.02-7702
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-10

CONDITIONS: Sports Physical Therapy
Keywords: Virtual reality; Wingate anaerobic test; Sports rehabilitation; performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evaluation Group (Other): Athletes are first assessed with the classic WAnT protocol in a laboratory environment with the same conditions at least 48 hours apart, then they perform the Wingate test (WAnT-VR) with the scenario integrated into the Oculus virtual reality goggles with the same protocol.
  Interventions: Device: Wingate Anaerobic Test with Virtual Reality

INTERVENTIONS:
Device: Wingate Anaerobic Test with Virtual Reality — Wingate Anaerobic Power Test Protocol, commonly used for assessing anaerobic capacity, involves a warm-up followed by testing. The warm-up includes 5 minutes of dynamic cycling, incorporating sprints. During the test, the athlete pedals at maximum effort for 30 seconds with added weight. Heart rate is monitored, and power output is measured every 5 seconds. Peak and average power values are calculated.
  This protocol will be gamified for VR goggles. The warm-up simulates cycling in a forest. Athletes sprint for 5 seconds every minute to escape a train, with prompts on the screen. The testing phase includes a simulated race, with athletes pedaling at maximum effort for 30 seconds to compete against rivals, signaled by flares and a countdown.
  Other Names: Wingate Anaerobic Test

SUMMARY:
Virtual reality (VR) is a technology utilizing three-dimensional graphical representations to immerse individuals in computer-generated environments, fostering engagement through visual, auditory, and tactile stimuli. VR applications offer enriched training environments, enhancing motor learning and autonomy, thus becoming integral in rehabilitation programs. Recent research underscores VR's efficacy in improving functional abilities across various conditions, including upper and lower limb disorders, balance, and cognitive impairments. Additionally, VR-based interventions demonstrate superiority over traditional methods in pain management, kinesiophobia prevention, and gait enhancement, particularly in conditions like cerebral palsy. The advantages of VR in therapy include its entertainment value, detailed performance feedback, simplicity, cost-effectiveness, and promotion of social interaction and cognitive function.

In sports, precise anaerobic assessment is crucial, especially for athletes engaging in high-intensity activities like sprinting and jumping. The 30-second Wingate Anaerobic Test (WAnT) is widely regarded as the gold standard for assessing anaerobic power, measuring peak power, average power, and fatigue index. External stimuli, such as verbal feedback and motivational guidance, influence test performance significantly, as evidenced by studies showing increased peak power and speed in athletes. Music has also been shown to enhance exercise performance, possibly through physiological synchronization with movement.

Integrating VR scenarios into assessment methods, such as the WAnT, may improve reproducibility and standardization by eliminating evaluator biases and ensuring consistent feedback levels. This study aims to explore the feasibility and efficacy of using VR-integrated WAnT in athletes, comparing its effects on performance to traditional applications.

DETAILED DESCRIPTION:
Virtual reality (VR) is defined as a three-dimensional graphical representation created by imaging technologies, where people are virtually present and real and imaginary environments are computer-generated. Applications that incorporate VR provide training in stimulating and enriched environments using visual, auditory, and tactile inputs. The virtual environment provides feedback to enhance motor learning and allows individuals to safely explore their environment independently by increasing their sense of autonomy in high-intensity training protocols. The effect of VR can be strong enough to allow participants to respond realistically. Participants' behavior can be altered as if they were exposed to a real-life scenario. Furthermore, being inside an avatar, where the virtual body feels like one's own, creates the perception that an action of the avatar is intended by the participant in their own brain.

In recent years, thanks to the advantages and possibilities offered by VR technologies, it has been widely used as an alternative rehabilitation program. It can improve functional abilities, such as repetition of specific tasks, in various rehabilitation patients. Literature has shown its benefits for upper and lower limb disorders, balance gait, and cognitive disorders. VR-based isokinetic training was found more effective than traditional exercise for pain management and preventing kinesiophobia. VR-based treadmill training in children with cerebral palsy has been shown to contribute more to gait quality, muscle strength gains, and the development of balance skills than classical treadmill training. The incorporation of VR applications into treatment programs has many advantages in use, such as reducing space and time dependency through entertainment and motivation, providing detailed feedback on performance, being simple, inexpensive, and reliable, allowing multiple repetitions of activities, stimulating motor learning and cortical plasticity, providing social interaction and supporting cognitive function.

The use of fast, high-intensity activities such as sprinting and jumping in sports makes accurate anaerobic assessment essential, particularly in athletes. Although many different methods/tests have been proposed for the measurement of anaerobic components, the 30-second Wingate Anaerobic Test (WAnT) is considered to be the gold standard. The WAnT is a maximal intensity cycle ergometer test developed in the 1970s. The commonly accepted performance components of the WAnT are peak power, average power, and fatigue index. Peak power is defined as the highest mechanical power achieved during the test in any 5-second period and is taken as the average power. Average power is the average power maintained over a 6x5 second period. The fatigue index is expressed as a percentage of the amount of drop in peak power during the test. The sum of these three components of power is considered to be an objective indicator of the anaerobic power of the athlete.

It is known that the visual, auditory, and tactile inputs provided externally to the individual during physiotherapy assessment enhance the individual's test performance and allow the test to be completed with maximum participation. Verbal feedback provided to the athlete showed an increase in the athlete's peak power and speed in the assessed upper body region in a study conducted on an elite group of athletes consisting of rugby players. This suggests that motivational guidance such as feedback or verbal encouragement given to the patient or sports person during the assessment may positively or negatively affect the assessment result. When a high level of performance is expected, external stimuli such as musical stimuli play a very important role in performance activation. Heart rate, respiratory rate, movement rate, and pulse rate tend to synchronize with the rhythm of the music. There is evidence in the literature that listening to music during WAnT can physiologically improve relative anaerobic exercise performance, although the reasons for this are speculative.

It suggests that assessment methods that include VR-integrated scenarios and provide auditory and visual feedback may be useful in terms of reproducibility by eliminating the differences between evaluators and ensuring that the verbal-auditory feedback given to participants during the assessment is at the same level. Our study aimed to investigate the applicability of goggle-integrated WAnT with virtual reality-based scenarios in athletes, evaluating the effect and difference of WAnT on performance compared to classical applications.

ELIGIBILITY:
Inclusion Criteria:

* To volunteer for the study and be between 18 and 25 years of age.
* To have successfully completed the classic Wingate test in previous periods

Exclusion Criteria:

* History of hospitalization for more than two weeks for any reason in the last three months,
* History of acute illness or injury during the study period
* Athletes who have not participated in training during the last two weeks will be excluded.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-14 (Actual)

PRIMARY OUTCOMES:
Wingate Anaerobic Test | for 30 seconds during testing
  The Wingate Anaerobic Test will be used as a tool to measure both muscular strength and anaerobic capacity in a 30-second time frame.

SECONDARY OUTCOMES:
System Usability Scale (SUS) | immediately after the Wingate Anaerobic Test with Virtual Reality
  SUS is a Likert scale. It is often assumed that a Likert scale is simply one based on forced choice questions, where a statement is made and the respondent then indicates the degree of agreement or disagreement with the statement on a 5 point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Bayram GA, Sahin GE, Yilmaz G, Tayboga UI, Celik AG, Yildirim Y, Saribas PK, Tarakci D. Integration of the wingate anaerobic test into a virtual reality- based evaluation system. BMC Sports Sci Med Rehabil. 2025 Jul 2;17(1):163. doi: 10.1186/s13102-025-01220-4. PMID 40605090